CLINICAL TRIAL: NCT06296407
Title: Integrated Psychophysical Analysis of Adolescent Patients With Obesity and Efficacy of the Respiratory Approach in Promoting the Condition of Psychophysical Well-being and the Performance of Physical Activity
Brief Title: Psychophysical Analysis of Adolescent Patients With Obesity and Efficacy of the Respiratory Approach (PSICOFISADOLOB).
Acronym: PSICOFISADOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 01C319
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Obesity, Childhood
Keywords: Obesity; Respiration; Physical activity; Psychophysical weel-being
MeSH Terms: conditions — Pediatric Obesity; Obesity; Respiratory Aspiration; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory exercises (Experimental): Males and females with obesity on standard metabolic integrated rehabilitation protocol + respiratory exercises
  Interventions: Other: Standard metabolic integrated rehabilitation protocol + respiratory exercises - duration 3 weeks
- Control (Active Comparator): Males and females with obesity on standard metabolic integrated rehabilitation protocol
  Interventions: Other: Standard metabolic integrated rehabilitation protocol - duration 3 weeks

INTERVENTIONS:
Other: Standard metabolic integrated rehabilitation protocol - duration 3 weeks — Standard metabolic integrated rehabilitation protocol
  Arms: Control
Other: Standard metabolic integrated rehabilitation protocol + respiratory exercises - duration 3 weeks — Standard metabolic integrated rehabilitation protocol + respiratory exercises (12 sessions [5 sessions/week for 3 weeks])
  Arms: Respiratory exercises

SUMMARY:
Specifically, the project aims to pursue the following objectives:

1. To evaluate in male and female adolescents with obesity the interaction between different psycho-body aspects such as respiration - posture - self-perception and affectivity and tolerance to physical exercise;
2. To evaluate in a subgroup of male and female adolescents the effectiveness of exercises aimed at respiratory muscles and of respiratory consciousness on the parameters above indicated and on their interaction.

The final objective of this project is to define and propose "take home" specific respiratory exercises to promote greater body awareness and a condition of psychophysical well-being stable over time, creating a condition that can favor further interventions on obesity. Finally, the project aims to build solid scientific bases to insert respiratory exercise among the intervention guidelines to prevent and reduce obesity, particularly youth obesity.

DETAILED DESCRIPTION:
Objectives:

Specifically, the project aims to pursue the following objectives:

1. To evaluate in male and female adolescents with obesity the interaction between different psycho-body aspects such as respiration - posture - self-perception and affectivity and tolerance to physical exercise;
2. To evaluate in a subgroup of male and female adolescents the effectiveness of exercises aimed at respiratory muscles and of respiratory consciousness on the parameters above indicated and on their interaction.

The final objective of this project is to define and propose "take home" specific respiratory exercises to promote greater body awareness and a condition of psychophysical well-being stable over time, creating a condition that can favor further interventions on obesity. Finally, the project aims to build solid scientific bases to insert respiratory exercise among the intervention guidelines to prevent and reduce obesity, particularly youth obesity. Material and Methods:

Participants:

24 males and females with obesity, aged between 12 and 18 years enrolled at the Division of Auxologia, Hospital San Giuseppe, Istituto Auxologico Italiano, IRCCS, Piancavallo (VB), Italy.

The participants are subdivided randomly into two subgroups: i. one control group (12 male and female adolescents) follows the standard metabolic integrated rehabilitation protocol and ii. an experimental group (12 male and female adolescents) who, in addition to the standard protocol, performs 12 sessions (5 sessions/week for 3 weeks) of 30 minutes each of respiratory exercises. The exercise definition are based on recent studies performed on obese patients (Batrakoulis 2022 a-b; Calcaterra et al., 2013-2014) and on different patient populations where the respiratory dysfunction is a primary or secondary pathology component (Bernardi et al., 2002). All the exercises are adapted to the examined population and guided and monitored by expert staff.

ELIGIBILITY:
Inclusion Criteria:

* BMI standard deviation score (SDS) > 2;
* absence of structured programs of physical activity (regular activity for more than 120min/week) for the 6 months before the study;
* absence of signs/symptoms related to cardiovascular, respiratory, gastrointestinal, skeletal-muscle pathologies contraindicated for the test execution

Exclusion Criteria:

* BMI standard deviation score (SDS) < 2;
* presence of structured programs of physical activity (regular activity for more than 120min/week) for the 6 months before the study;
* presence of signs/symptoms related to cardiovascular, respiratory, gastrointestinal, skeletal-muscle pathologies contraindicated for the test execution

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Fat mass | At baseline and after 3 weeks of intervention
  Assessed by tetrapolar impedance
Fat-free mass | At baseline and after 3 weeks of intervention
  Assessed by tetrapolar impedance
Maximal Inspiratory Pressure | At baseline and after 3 weeks of intervention
  Assessed by metabolimeter
Maximal Expiratory Pressure | At baseline and after 3 weeks of intervention
  Assessed by metabolimeter
Interoceptive awareness | At baseline and after 3 weeks of intervention
  Assessed by Multidimensional Assessment of Interoceptive Awareness Scale, with a self-report survey composed of 32 items with a Likert scale composed of 5 points scale

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Site Piancavallo, Oggebbio, Verbania, Italy